CLINICAL TRIAL: NCT04445025
Title: The Effect of Elagolix in Comparison to Leuprolide Acetate on in Vitro Fertilization (IVF) Cycle Outcomes After a Transfer of Euploid Embryos to Patients With Surgically Diagnosed Endometriosis: A Pilot Trial
Brief Title: Comparison Elagolix vs Depot Leuprolide Prior to Frozen Embryo Transfers in Patients With Endometriosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Colorado Center for Reproductive Medicine (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Eric Surrey, M.D., Medical Director, Colorado Center for Reproductive Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elagolix
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Infertility; Endometriosis
MeSH Terms: conditions — Infertility; Endometriosis | interventions — elagolix; Leuprolide

STUDY DESIGN:
Intervention Model Description: Test group will receive Elagolix 60 days prior to initiating frozen embryo transfer preparation.
  Control group will receive depot leuprolide twice (once every 28 days) prior to initiation frozen embryo transfer preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Subjects will receive the medication elagolix
  Interventions: Drug: Elagolix 200 MG; Diagnostic Test: Lab work
- Control group (Active Comparator): Subjects will receive leuprolide acetate
  Interventions: Drug: Leuprolide Acetate 3.75 MG/ML; Diagnostic Test: Lab work

INTERVENTIONS:
Drug: Elagolix 200 MG — Elagolix 200mg twice daily orally for 60 days prior to beginning frozen embryo transfer preparation
  Arms: Test group
Drug: Leuprolide Acetate 3.75 MG/ML — Leuprolide Acetate intramuscularly every 28 days (twice) prior to beginning frozen embryo transfer preparation
  Arms: Control group
Diagnostic Test: Lab work — Serum follicle stimulating hormone (FSH), estradiol, luteinizing hormone (LH), progesterone, human chorionic gonadotropin (hCG), serum for microarray analysis, complete blood count, and chemistry panel with liver functions levels will be drawn via blood draw

SUMMARY:
Patients who have been previously surgically diagnosed with endometriosis and have embryos predicted to be euploid after in vitro fertilization will be divided into 2 groups via randomization. The test group will receive Elagolix for 60 days prior to starting frozen embryo transfer preparation. The control group will be given leuprolide acetate every 28 days x 2 prior to starting the frozen embryo transfer preparation.

Comparative implantation rates between two groups of patients will be evaluated

DETAILED DESCRIPTION:
1. Baseline visit prior to initiation of IVF cycle:

   Review nature of study, confirm surgical diagnosis of endometriosis, obtain informed consent, confirm absence of exclusion criteria
2. Standard IVF and preimplantation genetic screening (prior to study entry):

   Subjects will undergo standard ovarian stimulation, monitoring (serum and ultrasound), oocyte aspiration, in vitro fertilization (IVF), intracytoplasmic sperm injection (ICSI), embryo culture to the blastocyst stage of development, trophectoderm biopsy, comprehensive chromosomal screening of embryos (CCS) and embryo vitrification as per protocols of CCRM and as determined by the primary CCRM physician.
3. Initial study entry visit performed within 4 weeks of initial medication administration after confirmation of presence of euploid embryo(s): Complete blood count, chemistry, renal and liver function panels. Computer generated randomization Obtain serum sample for micro RNA evaluation (results will not impact treatment and will only be analyzed retrospectively) Cycle Day2-4 serum FSH, estradiol, LH, progesterone, hCG level and transvaginal ultrasound examination to evaluate endometrial lining and the presence/absence of ovarian cysts All patients will be instructed to avoid pregnancy through use of barrier contraception while on study drug
4. Initial dosing Once screening evaluation has been cleared by the investigator, subject will be administered Lupron Depot 3.75 mg intramuscularly on cycle day 2-6 or will self-administer elagolix 200 mg orally twice daily beginning 2-6
5. Week 4 (30 days after initial dosing) Subjects will have repeat FSH, estradiol, LH, progesterone, and hCG levels drawn Subjects will be interviewed by study coordinator regarding presence or absence adverse outcomes/side effects including incidence and severity of hot flushes, vaginal bleeding, headache, nausea and vomiting Unless subject wishes to discontinue trial or is experiencing significant adverse events necessitating drop-out, patients in Lupron group will receive a second dose of Lupron Depot 3.75 mg intramuscularly and those in the elagolix dose will continue 200 mg twice daily oral dosing for an additional 30 days which will be dispensed at this visit
6. Week 8 (60 days after initial dosing) Subjects will have repeat FSH, estradiol, LH, progesterone and hCG levels as well as CBC and chem panel including liver function tests drawn Serum sample will be obtained for follow-up microarray analysis Transvaginal ultrasound examination will be performed to evaluate endometrial thickness and presence/absence of ovarian cysts Interview with study coordinator regarding presence/absence of adverse events/ side effects as described above
7. First menses after completion of study drug/ Endometrial preparation for embryo transfer Initiation of standard endometrial preparation with exogenous trans-dermal estradiol in conjunction with oral and/or intramuscular preparations per standard CCRM protocols and as determined by the primary physician to achieve an endometrial thickness of 7.0-15.0 mm with a trilaminar pattern. Standard monitoring with serial ultrasound examination and assessment of serial estradiol, LH and progesterone levels will be performed per CCRM protocols. Once appropriate endometrial development has been achieved after a minimum of 10 days of preparation, both intravaginal and intramuscular progesterone will be added to the estradiol with planned embryo transfer on the sixth day of progesterone administration
8. Embryo transfer Vitrified euploid embryo(s) selected for transfer will be warmed on the day of transfer which will be performed under ultrasound guidance using standard CCRM protocols. No more than 2 euploid embryos may be transferred and all patients will be encouraged to undergo a single transfer. Indication for a two embryo transfer will be documented. Best quality embryo(s) will be transferred preferentially choosing day 5 euploid blastocysts over day 6 or 7 euploid blastocysts. Embryos will be graded using the classification system of Gardner et al. (see reference section)
9. Luteal support Subjects will receive standard luteal support with both injectable and intravaginal progesterone with doses adjusted per CCRM guidelines.
10. Pregnancy diagnosis and monitoring Subjects will have an initial serum hCG level obtained 9 days after embryo transfer in their local clinic. Estradiol and progesterone levels will also be measured if hCG is positive. Repeat hCG level will obtained two days after the first level if the first level was positive. First pregnancy ultrasound will be obtained 2-2.5 weeks after initial positive hCG level unless there is a clinical indication for an earlier evaluation. If all is normal with first pregnancy ultrasound examination, a second ultrasound examination to evaluate pregnancy will be performed 2-2.5 weeks thereafter unless clinical circumstances require earlier evaluation. Progesterone and estradiol supplementation will typically be tapered using CCRM guidelines beginning at 10 weeks of pregnancy and be discontinued entirely no later than the end of the 13th week of pregnancy. Subjects will be referred to their primary obstetricians after the second pregnancy ultrasound examination at 8 weeks of pregnancy
11. Pregnancy outcome data collection The outcomes of all pregnancies shall be obtained from the patient and recorded. If live birth, all data required by Center for Disease Control will be collected including gestational age, birth weight, immediately diagnosed anomalies and pregnancy complications. The gestational age, management, and pathology reports (if available) from pregnancy loss, ectopic pregnancy and still birth shall also be collected.

Any pregnancies that occur while on study drugs or which occur after completion of the drugs but prior to embryo transfer will be recorded and monitored in the same fashion as described above

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of infertility who are candidate for IVF
2. Surgical diagnosis of endometriosis within 10 years of study entry
3. Willing to sign/give informed consent and adhere to parameters of study
4. Normal endometrial cavity as diagnosed by 3D ultrasound and office hysteroscopy examinations at baseline or after correction of underlying clinically relevant cavity abnormalities
5. Day 2-4 serum FSH level ≤ 12 mIu/mL and/or random serum AMH level ≥ 0.9 ng/mL and/or antral follicular phase follicle count obtained by trans-vaginal ultrasound examination ≥ 5
6. No contraindication to GnRH agonist or GnRH antagonist use
7. No prolonged use of GnRH agonist or antagonist (> 30 consecutive days) or other treatment for endometriosis within 4 months of study entry
8. Have at least one euploid embryo available for transfer
9. Agrees to transfer best quality embryo as determined by CCRM physician and embryology team
10. Regular menses ranging from 22-36 days
11. Agrees to use barrier contraception throughout GnRH agonist or antagonist administration
12. No evidence of untreated hydrosalpinx

Exclusion Criteria:

1. Age <21 or > 42 years at time of initiation of IVF cycle
2. Day 2-4 FSH level >12 mIu/mL or random serum AMH level <1.0 ng/mL and antral follicle count obtained by trans-vaginal ultrasound examination < 5
3. Planned use of donor oocytes or embryos
4. Planned use of gestational carrier
5. Use of GnRH agonist, GnRH antagonist or other approved medical therapy for endometriosis (with the exception of combination contraceptives) for > 30 consecutive days prior to study entry
6. Unwilling to abide by study parameters or sign informed consent
7. No documentation of surgical diagnosis of endometriosis with study timeline (10 years of study entry)
8. Absence of embryos predicted to be euploid available for transfer (embryos with no results may not be included in transfer)
9. Prior adverse reaction to any GnRH agonist or antagonist
10. Uncorrected or uncorrectable clinically relevant uterine cavity abnormalities or hydrosalpinx
11. Acute or chronic renal, pulmonary, hepatic, or cardiac disease
12. Prior diagnosis of pituitary adenoma or any other intracranial lesion
13. Menstrual cycles outside the range of inclusion criteria
14. Diagnosis of polycystic ovary syndrome (PCOS)
15. Pregnancy prior to study initiation or initiation of endometrial preparation for embryo transfer.
16. Undiagnosed vaginal bleeding
17. Clinically relevant adenomyosis as diagnosed by baseline 3D ultrasound exam (and/or MRI if felt to be appropriate)
18. Bipolar disorder, history of suicidal ideation, any other psychiatric disorder requiring lithium or anti-psychotic medications

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Implantation Rates | 2-3 weeks after initial positive pregnancy test (approx 14-15 weeks post initiation of treatment)
  Implantation rates of both groups will be compared (defined as number of intrauterine gestational sacs with visible cardiac activity noted on ultrasound examination performed 2-3 weeks after initial positive pregnancy test)

SECONDARY OUTCOMES:
Comparison of Biochemical pregnancy rates | 2-3 weeks after initial positive pregnancy test (approx 14-15 weeks post initiation of treatment)
  Comparative biochemical pregnancy rates (positive pregnancy tests with no evidence of intrauterine gestational sac noted at ultrasound performed 2-3 weeks after initial positive pregnancy test) per embryo transfer
Comparison of hormone levels between the two groups | 4 weeks and 8 weeks after initiation of treatment
  FSH, LH, Estradiol, progesterone will compared after 4 weeks and 8 weeks of initiation of treatment
Comparison of live birth rates and pregnancy loss rates | 10-11 months after initiation of treatment
  At the end of the pregnancy. Live birth rates and pregnancy loss rates will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Eric Surrey, MD, Principal Investigator — Colorado Center for Reproductive Medicine
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosar E, Mamillapalli R, Ersoy GS, Cho S, Seifer B, Taylor HS. Serum microRNAs as diagnostic markers of endometriosis: a comprehensive array-based analysis. Fertil Steril. 2016 Aug;106(2):402-9. doi: 10.1016/j.fertnstert.2016.04.013. Epub 2016 May 11. PMID 27179784
- [Background] Schoolcraft WB, Treff NR, Stevens JM, Ferry K, Katz-Jaffe M, Scott RT Jr. Live birth outcome with trophectoderm biopsy, blastocyst vitrification, and single-nucleotide polymorphism microarray-based comprehensive chromosome screening in infertile patients. Fertil Steril. 2011 Sep;96(3):638-40. doi: 10.1016/j.fertnstert.2011.06.049. Epub 2011 Jul 23. PMID 21782169
- [Background] Surrey ES, Minjarez DA, Schoolcraft WB. The incidence of aberrant endometrial alphavbeta(3) vitronectin expression in a high risk infertility population: could prolonged GnRH agonist therapy play a role? J Assist Reprod Genet. 2007 Nov;24(11):553-6. doi: 10.1007/s10815-007-9164-3. Epub 2007 Nov 17. PMID 18026832
- [Background] Taylor HS, Giudice LC, Lessey BA, Abrao MS, Kotarski J, Archer DF, Diamond MP, Surrey E, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Rowan JP, Duan WR, Ng J, Schwefel B, Thomas JW, Jain RI, Chwalisz K. Treatment of Endometriosis-Associated Pain with Elagolix, an Oral GnRH Antagonist. N Engl J Med. 2017 Jul 6;377(1):28-40. doi: 10.1056/NEJMoa1700089. Epub 2017 May 19. PMID 28525302
- [Background] Surrey ES, Katz-Jaffe M, Kondapalli LV, Gustofson RL, Schoolcraft WB. GnRH agonist administration prior to embryo transfer in freeze-all cycles of patients with endometriosis or aberrant endometrial integrin expression. Reprod Biomed Online. 2017 Aug;35(2):145-151. doi: 10.1016/j.rbmo.2017.05.004. Epub 2017 May 17. PMID 28601378
- [Background] Gardner DK, Surrey E, Minjarez D, Leitz A, Stevens J, Schoolcraft WB. Single blastocyst transfer: a prospective randomized trial. Fertil Steril. 2004 Mar;81(3):551-5. doi: 10.1016/j.fertnstert.2003.07.023. PMID 15037401
- [Background] Sallam HN, Garcia-Velasco JA, Dias S, Arici A. Long-term pituitary down-regulation before in vitro fertilization (IVF) for women with endometriosis. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD004635. doi: 10.1002/14651858.CD004635.pub2. PMID 16437491
- [Result] Surrey ES, Silverberg KM, Surrey MW, Schoolcraft WB. Effect of prolonged gonadotropin-releasing hormone agonist therapy on the outcome of in vitro fertilization-embryo transfer in patients with endometriosis. Fertil Steril. 2002 Oct;78(4):699-704. doi: 10.1016/s0015-0282(02)03373-3. PMID 12372443